CLINICAL TRIAL: NCT06621277
Title: JUMP_START - Optimization of Care for Young Cancer Patients with Gastrointestinal Tumors
Acronym: JUMP_START
Status: Recruiting | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Bruno Christian Köhler, Principal Investigator, University Hospital Heidelberg
Other Study IDs: NCT_GI_BCK_02; AIO-LQ-0323ass (Other: AIO Germany)
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Gastrointestinal Cancer
Keywords: Quality of Life; gastrointestinal tumors
MeSH Terms: conditions — Gastrointestinal Neoplasms; Digestive System Neoplasms | interventions — Clinical Trials, Phase II as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Individuals received a GI tumor diagnosis > 50 years
  Interventions: Other: No intervention
- Individuals received a GI tumor diagnosis ≤ 50 years
  Interventions: Other: Tailored counseling programs (Phase 2)

INTERVENTIONS:
Other: No intervention — No intervention
  Groups: Individuals received a GI tumor diagnosis > 50 years
Other: Tailored counseling programs (Phase 2) — Optimized care services and tailored counseling programs for young patients with GI tumors at the Heidelberg University Hospital (Phase 2)
  Groups: Individuals received a GI tumor diagnosis ≤ 50 years

SUMMARY:
JUMP_START aims to assess the needs of individuals aged ≤ 50 years with gastrointestinal (GI) tumors and implement a tailored support and counseling program at the University Hospital Heidelberg and the National Center for Tumor Diseases (NCT).

In phase 1A, 12-15 individuals aged ≤ 50 years with GI tumors will be interviewed via telephone using semi-structured interviews to obstain a detailed understanding of the life situation, the burdens, and the care situation within the structures of the NCT Heidelberg.

In phase 1B, the care networks of young patients with GI tumors beyond the NCT, including the analysis of changes and important access routes/possible gatekeepers, will be explored using so-called ego-centered network analyses, in comparison with patients who received a GI tumor diagnosis after the age of 50.

In response to the results of phase 1A and 1B, the care services for young patients with GI tumors will be optimized, and tailored counseling programs will be developed in phase 2.

These project phases will be accompanied by Quality of Life assessments using European Organisation for Research and Treatment of Cancer (EORTC) questionnaires. All patients with GI tumors (regardless of potential inclusion in phase 1A or 1B) will receive the EORTC questionnaires once. In phase 2, Quality of Life will be assessed every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged ≥ 18 and ≤ 50 years receiving treatment for a GI tumor at the Heidelberg University Hospital
* Sufficient knowledge of the German language
* Capable of providing informed consent
* Additional recruitment for Phase 1B and Quality of Life assessments: Patients with GI tumor aged ≥ 51 years

Exclusion Criteria:

* Individuals with a GI tumor diagnosis after the age of 50 (except in Phase 1B and for Quality of Life assessments)
* Individuals with a GI tumor diagnosis under the age of 18
* Lack of capacity to consent and/or absence of informed consent
* Insufficient knowledge of the German language
* Severe cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with a GI tumor diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Quality of Life at two years | Baseline, 6; 12; 18, and 24 months
  Changes in Quality of Life in patients aged ≤ 50 years with a GI tumor diagnosis who are using optimized counseling programs will be measured using EORTC questionnaires (e.g. EORTC-QLQ C30, EORTC QLQ-CR29, EORTC LMC21, EORTC HCC18, EORTC QLQ-OG25). Scores will be categorized into functional and symptom scales (0-100 range) following the EORTC Scoring Manual. For Functional scales and Global QoL: Higher scores indicate better functioning or better QoL. For Symptom scales: Higher scores indicate greater symptom burden.

OTHER OUTCOMES:
Differences in Quality of Life between patients aged ≤ 50 years and > 50 years | Once at baseline, after enrollment
  Differences in Quality of Life in patients aged ≤ 50 years and > 50 years with a GI tumor diagnosis will be measured using EORTC questionnaires (e.g. EORTC-QLQ C30, EORTC QLQ-CR29, EORTC LMC21, EORTC HCC18, EORTC QLQ-OG25). Scores will be categorized into functional and symptom scales (0-100 range) following the EORTC Scoring Manual. For Functional scales and Global QoL: Higher scores indicate better functioning or better QoL. For Symptom scales: Higher scores indicate greater symptom burden.

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Tumor Diseases (NCT) Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared for scientific collaborations after agreement with PI.